CLINICAL TRIAL: NCT01535014
Title: Multicentric Double-blind Placebo-controlled Randomized Parallel-group Clinical Trial of Safety and Efficacy of Various Dosage Schedules for Dietressa Drug in Treatment of Obese Patients
Brief Title: Clinical Trial of Safety and Efficacy of Various Dosage Schedules for Dietressa Drug in Treatment of Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-DI-002
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Dietressa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dietressa (2 tablets 3 times daily) for 24 weeks (Experimental): Patients with Body Mass Index 30.0-34.9 (kg/m2) without previous anti-obesity treatment received Dietressa (2 tablets 3 times daily) for 24 weeks.
  Interventions: Drug: Dietressa
- Dietressa (1 tablet 6 times daily) for 24 weeks (Experimental): Patients with Body Mass Index 30.0-34.9 (kg/m2) without previous anti-obesity treatment received Dietressa (1 tablet 6 times daily) for 24 weeks.
  Interventions: Drug: Dietressa
- Placebo (2 tablets 3 times daily) (Placebo Comparator): Patients with Body Mass Index 30.0-34.9 (kg/m2) without previous anti-obesity treatment received Placebo (2 tablets 3 times daily) for 24 weeks.
  Interventions: Drug: Placebo
- Placebo (1 tablet 6 times daily) (Placebo Comparator): Patients with Body Mass Index 30.0-34.9 (kg/m2) without previous anti-obesity treatment received Placebo (1 tablet 6 times daily) for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dietressa — Comparison of different dosages (frequency) of drug
  Arms: Dietressa (1 tablet 6 times daily) for 24 weeks; Dietressa (2 tablets 3 times daily) for 24 weeks
Drug: Placebo — Placebo either (2 tablets 3 times daily) or
  (1 tablet 6 times daily)
  Arms: Placebo (1 tablet 6 times daily); Placebo (2 tablets 3 times daily)

SUMMARY:
The purpose of this study is:

* To assess safety of Dietressa in the dose of 6 tablets daily within 24 weeks in treatment of obese patients.
* To assess clinical efficacy of Dietressa in the dose of 6 tablets daily within 24 weeks of therapy in reducing body weight in obese patients.
* To compare clinical efficacy of two dosage patterns for Dietressa (1 tablet 6 times daily and 2 tablets 3 times daily) within 24 weeks in treatment of obese patients.

DETAILED DESCRIPTION:
In general, patients will be observed during 24 weeks of trial.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient subjects with BMI 30,0-34,9 kg/m2.
2. Male or female subjects aged 18 to 65 inclusive.
3. Use of and compliance with contraception methods by patients of reproductive age, of both sexes.
4. Presence of the patient's information sheet (informed consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Symptomatic (secondary) obesity:

   * with established genetic defect (including as a part of known genetic syndromes affecting multiple organs): Prader-Willi syndrome, Alstrom's syndrome, Laurence-Moon-Biedl syndrome, Dercum's syndrome etc.
   * cerebral (adiposogenital dystrophy, Babinski-Frohlich syndrome): brain tumors; dissemination of systemic lesions, infectious diseases; against mental diseases.
   * endocrine: hypothyroid; hypoovarial; pituitary-hypothalamic disorders; adrenopathy.
   * iatrogenic (caused by drug administration, namely, insulin, glucocorticosteroids, neuroleptics etc.).
2. Compliance with a diet prescribed and monitored by the doctor to reduce body weight within 6 months before enrollment.
3. Participation in the lifestyle modification program within 6 months before enrollment.
4. Patients who quit smoking within 6 months before enrollment, or intending to quit smoking during the period of participation in the trial, as well as intending to begin smoking during the trial.
5. Uncontrolled arterial hypertension (patients with 1-3 degree AH, receiving no adequate antihypertensive therapy).
6. Type 1 and 2 diabetes mellitus.
7. Edema syndrome with various etiology (chronic cardiac failure, nephrotic syndrome, hepatic cirrhosis).
8. Circulatory failure, IIА degree and above.
9. Decompensated cardiovascular disease, liver, kidney or gastrointestinal tract disease, metabolic, respiratory, endocrine, hematologic disease, peripheral vessel disease or another medical state. Oncological disease.
10. Diseases and states, which, in the investigator's opinion, may prevent the patient from participating in the trial.
11. Past history of bulimia / non-drug abepithymia.
12. Past history of any bariatric surgeries.
13. Lipoplasty underwent less then 1 year prior to screening visit, or cavitary surgery less then 6 months prior to screening visit.
14. Surgeries scheduled within 6 months.
15. Allergy to/intolerance of any of the drug components used during treatment.
16. Malabsorption syndrome, including congenial or acquired lactase or another disaccharidase insufficiency.
17. Administration of drugs specified as "Prohibited concomitant therapy", within 6 months before enrollment.
18. Pregnancy, breast-feeding, unwillingness to comply with contraception methods during the trial and within 30 days after completion of participation in the trial.
19. Drug and alcohol consumption (over 2 alc. units daily), mental diseases. Legal incapacity or limited legal capacity.

21. Patients, who, in the investigator's opinion, will fail to observe the requirements during the trial or adhere to the studied drug administration procedure.

22. Participation in other clinical trials within 3 months before enrolment in this trial.

23. Presence of other factors, complicating the patient's participation in the trial (e.g., planned lengthy business and other trips). 24. A patient is a part of the center's research staff, taking a direct part in the trial, or an immediate family member of the investigator. Immediate family members are defined as spouses, parents, children or siblings, regardless of whether full blood or adopted.

25. The patient is employed with Scientific Production Firm Materia Medica Holding LLC, i.e. is the company's employee, part-time employee under contract, or appointed official in charge of the trial, or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - The State Educational institution of High Professional Training Kuban State Medical University of Ministry of Health Care and Social Development of the Russian Federation, Department of Clinical Pharmacology, Krasnodar
  - The State Educational institution of High Professional Training I.M. Sechenov First Moscow State Medical University of Ministry of Health Care and Social Development of the Russian Federation, Endocrinology Faculty, Moscow
  - The State Budget Health Care institution of Moscow the City Clinical Hospital No. 11 of the Administration of Health Care of Moscow City, Moscow
  - Municipal Medical and Preventive institution "City Clinical Hospital No.10", Nizhny Novgorod
  - The State Budget Health Care institution of Nizhegorodskyi Region "Nizhegorodskaya Regional Clinical Hospital n.a. N.A.Semashko", Nizhny Novgorod
  - The State Educational institution of High Professional Training "Rostov State Medical University" of Ministry of Health Care and Social Development of the Russian Federation, Department of Endocrinology, Rostov-on-Don
  - St. Petersburg State Health Care institution "Municipal Hospital No.6", Saint Petersburg
  - St. Petersburg State Health Care institution "Municipal Hospital No.77 of Nevsky District", The City Diabetes Center, Saint Petersburg
  - The Federal State Health Care institution L.G. Sokolov Memorial Hospital No. 122 of the FMBA (Federal Medical and Biological Agency)., Saint Petersburg
  - The State Educational institution of High Professional Training "St. Petersburg State Medical University n.a. I.P. Pavlov of the Federal Agency for Health Care and Social Development", Faculty Surgery Board, Saint Petersburg
  - The State Educational institution of High Professional Training "St. Petersburg State Medical University n.a. I.P. Pavlov of the Federal Agency for Health Care and Social Development", Therapy Faculty Board, Saint Petersburg
  - St. Petersburg state Health Care institution "Saint Venerable Martyr Elizaveta Municipal Hospital", Saint Petersburg
  - St. Petersburg State Health Care institution "Consultative and Diagnostic Center No. 85", Diabetes Center, Saint Petersburg
  - The State Educational institution of High Professional Training "Bashkirsky State Medical University" of the Federal Agency for Health Care and Social Development, Department of Endocrinology, Ufa
  - The State Educational institution of High Professional Training "Volgograd State Medical University" of Ministry of Health Care and Social Development of the Russian Federation, Volgograd
  - The State Health Care institution "Voronezh Regional Clinical Consultative & Diagnostic Center", Voronezh
  - The State Health Care institution of Yaroslavl Region the Clinical Hospital, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietressa 1: Dietressa: 1 tablet 6 times daily
- Dietressa 2: Dietressa: 2 tablets 3 times daily
- Placebo 3: Placebo: 1 tablet 6 times daily
- Placebo 4: Placebo: 2 tablets 3 times daily
Period: Overall Study
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Started | 210 | 200 | 50 | 33
Completed | 208 | 194 | 49 | 33
Not Completed | 2 | 6 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4 | Total
Number analyzed (Participants) | 208 | 194 | 49 | 33 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.1) | 42.4 (12.1) | 41.4 (10.3) | 42.8 (11.3) | 41.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 167 | 44 | 30 | 422
  Male | 27 | 27 | 5 | 3 | 62
Height [Mean (Standard Deviation); unit: centimeter] | 166.4 (8.3) | 165.1 (7.9) | 164.4 (6.7) | 164.9 (7.8) | 165.6 (8.0)
Weight [Mean (Standard Deviation); unit: kilogram] | 89.1 (10.6) | 87.5 (9.5) | 87.1 (7.7) | 86.1 (9.8) | 88.1 (9.9)
BMI [Mean (Standard Deviation); unit: kilogram/m^2] | 32.1 (1.4) | 32.0 (1.5) | 32.2 (1.5) | 31.6 (1.3) | 32.0 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Lose at Least 5 Percent of Baseline Body Weight After 24 Weeks of Treatment Weeks of Treatment
Time Frame: assessed after 24 weeks of treatment
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
percentage of participants | 49 | 48 | 33 | 21
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p = 0.04, Chi-squared
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p = 0.004, Chi-squared
Statistical Analysis 3: Comparison: Dietressa 1 vs Dietressa 2 vs Placebo 3 vs Placebo 4; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel

2. Primary Outcome: Average Body Weight Change After 24 Weeks of Treatment
Time Frame: assessed after 24 weeks of treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
kilogram | -4.4 (4.2) | -4.4 (4.4) | -3.0 (3.5) | -2.9 (2.8)
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p = 0.07, t-test, 2 sided

3. Primary Outcome: Average Relative Change in Body Weight After 24 Weeks of Treatment
Time Frame: assessed after 24 weeks of treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
percentage of body weight | -4.9 (4.7) | -4.9 (4.9) | -3.4 (4.2) | -3.4 (3.3)
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p = 0.07, t-test, 2 sided

4. Secondary Outcome: Percentage of Subjects With a Decrease in Body Weight by 5 or More Percent of Baseline Body Weight After 4, 8, 12, 16, 20 and 24 Weeks of Treatment
Time Frame: assessed after 4, 8, 12, 16, 20, and 24 weeks of treatment
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
percentage of participants
  4 weeks | 4 | 5 | 4 | 0
  8 weeks | 17 | 16 | 8 | 3
  12 weeks | 26 | 24 | 12 | 15
  16 weeks | 34 | 36 | 16 | 18
  20 weeks | 38 | 42 | 22 | 15
  24 weeks | 49 | 48 | 33 | 21
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p < 0.05, Chi-squared — For week 12, 16, 20, 24
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p < 0.05, Chi-squared — For week 16, 20, 24

5. Secondary Outcome: Average Relative Weight Change After 4, 8, 12, 16, 20 and 24 Weeks of Treatment
Time Frame: assessed after 4, 8, 12, 16, 20 and 24 weeks of treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
percentage of body weight
  4 weeks | -1.5 (1.8) | -1.4 (2.1) | -0.8 (2.1) | -0.8 (1.4)
  8 weeks | -2.5 (2.6) | -2.5 (2.7) | -1.3 (3.8) | -1.5 (1.9)
  12 weeks | -3.2 (3.1) | -3.3 (3.4) | -2.1 (3.2) | -2.2 (2.7)
  16 weeks | -3.9 (3.7) | -4.0 (3.9) | -2.8 (3.7) | -2.6 (2.8)
  20 weeks | -4.3 (4.1) | -4.5 (4.4) | -3.1 (4.0) | -2.8 (3.1)
  24 weeks | -4.9 (4.7) | -4.9 (4.9) | -3.4 (4.2) | -3.4 (3.3)
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p = 0.019, ANCOVA
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p = 0.043, ANCOVA

6. Secondary Outcome: Waist Hip Ratio After 4, 12 and 24 Weeks of Treatment
Time Frame: assessed after 4,12 and 24 weeks of treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: waist hip ratio
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
waist hip ratio
  0 week | 0.88 (0.08) | 0.89 (0.09) | 0.89 (0.07) | 0.86 (0.08)
  4 weeks | 0.88 (0.08) | 0.89 (0.09) | 0.88 (0.08) | 0.85 (0.08)
  12 weeks | 0.88 (0.08) | 0.88 (0.09) | 0.87 (0.08) | 0.85 (0.08)
  24 weeks | 0.87 (0.08) | 0.88 (0.09) | 0.87 (0.08) | 0.85 (0.08)
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; Test type: Superiority; p = 0.20, ANCOVA
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; Test type: Superiority; p = 0.75, ANCOVA

7. Secondary Outcome: Change in the Quality of Life According to the Data of SF-36 Health Status Survey Questionnaire (SF-36) After 4, 12 and 24 Weeks of Treatment
Description: 36 items of the questionnaire are grouped into eight subscales. The subscales are grouped in two scales: the "physical component of health" and "mental health component". The scores of each scale range between 0 and 100: the higher the score, the better the quality of life and the better the patient's health.
  The instruction is not given completely because of the large volume. For more information, see: Ware J.E., Snow K.K., Kosinski M., Gandek B. SF-36 Health Survey. Manual and interpretation guide //The Health Institute, New England Medical Center. Boston, Mass.-1993. In this instruction is explained how eight subscales are combined to compute a total score.
Time Frame: baseline, 4, 12 and 24 weeks
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Dietressa 1 | Dietressa 2 | Placebo 3 | Placebo 4
Number analyzed (Participants) | 208 | 194 | 49 | 33
scores on a scale
  0 week (mental) | 43.7 (9.5) | 43.4 (10.4) | 44.3 (9.5) | 47.5 (7.3)
  4 weeks (mental) | 46.4 (9.3) | 46.1 (9.8) | 49.0 (9.1) | 49.5 (8.0)
  12 weeks (mental) | 46.5 (9.3) | 46.6 (10.2) | 49.3 (6.3) | 49.0 (8.6)
  24 weeks (mental) | 48.3 (8.7) | 47.5 (9.2) | 50.6 (7.0) | 50.0 (8.6)
  0 week (physical) | 50.0 (7.9) | 49.5 (7.3) | 49.5 (7.3) | 50.7 (7.6)
  4 weeks (physical) | 51.2 (7.1) | 50.1 (6.8) | 51.0 (6.8) | 51.5 (6.9)
  12 weeks (physical) | 52.2 (6.4) | 50.8 (7.2) | 51.3 (5.9) | 50.7 (7.8)
  24 weeks (physical) | 52.4 (6.5) | 51.3 (6.9) | 51.7 (6.2) | 52.3 (6.2)
Statistical Analysis 1: Comparison: Dietressa 1 vs Placebo 3; SF-36 Mental Health Domain; Test type: Superiority; p = 0.02, ANCOVA
Statistical Analysis 2: Comparison: Dietressa 2 vs Placebo 4; SF-36 Mental Health Domain; Test type: Superiority; p = 0.63, ANCOVA
Statistical Analysis 3: Comparison: Dietressa 1 vs Placebo 3; SF-36 Physical Health Domain; Test type: Superiority; p = 0.60, ANCOVA
Statistical Analysis 4: Comparison: Dietressa 2 vs Placebo 4; SF-36 Physical Health Domain; Test type: Superiority; p = 0.98, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 12 months of therapy and 30 days after the end of the research
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=493, Safety Population)
Groups:
- Dietressa 1+2: Dietressa 1: 1 tablet 6 times daily; Dietressa 2: 2 tablets 3 times daily
- Placebo 3+4: Placebo 3: 1 tablet 6 times daily; Placebo 4: 2 tablets 3 times daily
Arm/Group | Dietressa 1+2 | Placebo 3+4
Serious Adverse Events (participants affected / at risk) | 3/410 | 0/83
Other Adverse Events (participants affected / at risk) | 160/410 | 33/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietressa 1+2 (N=410) | Placebo 3+4 (N=83)
Uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0
Pregnancy NOS (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0
Intervertebral disc sequestration (Musculoskeletal and connective tissue disorders) | 1 (3) | 0
Vertebral osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (4) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dietressa 1+2 (N=410) | Placebo 3+4 (N=83)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 3
iron-deficient anemia (Blood and lymphatic system disorders) | 1 | 0 — mild disease
Сoronary artery disease (Cardiac disorders) | 1 | 0
Complaints about palpitations, sweating (Cardiac disorders) | 0 | 1
Autoimmune thyroiditis. Subclinical hypothyroidism (Endocrine disorders) | 1 | 0
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Dentalgia (Gastrointestinal disorders) | 1 | 0
Epigastric burning (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 — nausea after taking the drug before eating
Heaviness in the right hypochondrium (Gastrointestinal disorders) | 1 | 0
Enzymatic insufficiency (Gastrointestinal disorders) | 1 | 0 — ulcerative disease
Сhronic gastritis (Gastrointestinal disorders) | 1 | 0 — acute exacerbation of a chronic disease
Frequent stool up to 3 times a day (Gastrointestinal disorders) | 1 | 0
intestinal obstruction (Gastrointestinal disorders) | 0 | 1
exacerbation of chronic pancreatitis (Gastrointestinal disorders) | 0 | 1
Pastosity of the shins (General disorders) | 1 | 0
Acroedema (General disorders) | 1 | 0
Increase of ability to work (General disorders) | 1 | 0
Thirst perception (General disorders) | 0 | 1 — drinks more fluids
Hepatitis (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Acute respiratory viral infection (Infections and infestations) | 12 | 4
Acute respiratory disease (Infections and infestations) | 3 | 0
Acute respiratory disease (Infections and infestations) | 1 | 0 — with tracheobronchitis
Acute bronchitis (Infections and infestations) | 4 | 0
Acute laryngitis (Infections and infestations) | 1 | 0
Acute rhinopharyngitis (Infections and infestations) | 2 | 2
Acute pharyngitis (Infections and infestations) | 1 | 1
Cold (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0
Ligamentous injury (Injury, poisoning and procedural complications) | 0 | 1 — 1st metacarpophalangeal right hand joint
Increase in arterial pressure (Investigations) | 2 | 1
LDL increase (Investigations) | 1 | 0
C-reactive protein increase (Investigations) | 1 | 0
Glucose level increase (Investigations) | 3 | 0
Total cholesterol increase (Investigations) | 1 | 0
HDL increase (Investigations) | 2 | 1
Erythrocyte sedimentation rate increase (Investigations) | 2 | 2
Lymphocytosis level increase (Investigations) | 1 | 0
ALT increase (Investigations) | 0 | 2
Basophilia (Investigations) | 0 | 1
Erytrocytosis (Investigations) | 0 | 2
Leukocytosis (Investigations) | 0 | 1
Monocytosis (Investigations) | 0 | 2
Thrombocytopenia (Investigations) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 11 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 — Feeling appetite suppressed, decreased feelings of hunger
Suppressing appetite (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 1
Suppressing appetite (Investigations) | 1 | 0 — Suppressing appetite, feeling of saturation, has become overeat
Hyperglycaemia fasting (Metabolism and nutrition disorders) | 3 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 2 | 1
Hypercholesteremia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 — for sweet food
Periodic strong desire to eat something (Metabolism and nutrition disorders) | 0 | 1
Dorsopathy of a spine (Musculoskeletal and connective tissue disorders) | 2 | 0
gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 — left
Stiffness in hands (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Right shoulder joint arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Left hip joint arthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Unpleasant sweetish taste in a mouth (Nervous system disorders) | 1 | 0
Vertebral radiculopathy with moderate musculo-tonic and pain syndrome (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 1
Clinical anxiety (Psychiatric disorders) | 4 | 0
Subclinical anxiety (Psychiatric disorders) | 32 | 6
Increased anxiety on a scale HADS (Psychiatric disorders) | 42 | 8
Mood changes: a tendency towards depression, aggressiveness (Psychiatric disorders) | 1 | 0
Subclinical depression (Psychiatric disorders) | 20 | 2
Clinical depression (Psychiatric disorders) | 6 | 0
Increased depression on a scale HADS (Psychiatric disorders) | 36 | 4
Exaggeratedly mood, unreasonable euphoria (Psychiatric disorders) | 1 | 0
Unpleasant smell of urine (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness and throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin rash (allergic reaction) (Skin and subcutaneous tissue disorders) | 1 | 0
Increased brittleness of nails (Skin and subcutaneous tissue disorders) | 1 | 1
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Xerosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertensic crisis (Vascular disorders) | 1 | 0
Hypotonia (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other